CLINICAL TRIAL: NCT03071952
Title: Assessment of AAIR Pacing Treatment for Heart Failure Patients With Chronotropic Incompetence
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: CI Study Phase II
Record Dates: First submitted 2016-09-08; First posted 2017-03-07 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Chronotropic Incompetence; Rate Response; Exercise Test
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to assess the clinical efficacy of AAIR (Atrial-paced Atrial-sensed Inhibitory Rate-Modulated) pacing treatment for heart failure (HF) patients with chronotropic incompetence (CI) in terms of exercise tolerance and quality of life. Specifically, the study will assess the changes in cardiac function associated with changes of physical exercise intensity and heart rate in AAIR pacing mode compared with AAI pacing mode.

DETAILED DESCRIPTION:
CI is the inability of the heart to increase its rate in response to increased physical activity or metabolic demand, leading to exercise intolerance and poor quality of life. Studies have demonstrated that patients with CI have a high risk of cardiac morbidity and mortality. Recent studies further demonstrate a high incidence of CI in patients with heart failure, which is also confirmed by CI in Heart Failure Study Phase I. However, clinical attention is often paid to heart failure symptoms instead CI-related symptom. Thus, patients with heart failure are often not tested for CI, even though the CI incidence is high in these patients. Moreover, such patients could gain significant improvements in exercise tolerance and quality of life once they get diagnosed followed by effective therapy for CI and long-term management.

This study is designed to establish clinical evidence that AAIR pacing is beneficial to treat CI-caused symptoms in heart failure patients, which will improve the life quality of such patients and further support the expansion of Brady therapy indications to the population of HF with CI in existing markets and also potential markets.

CI is rarely seen and has different definition among various animal species. It is impossible to use animals to get wanted data for AAIR pacing treatment to CI. Thus, a human clinical study is necessary. Furthermore, exercise testings, such as 6 minutes hall walk (6MHW) and treadmill, allow objective evaluation of exercise capacity and exertional symptoms, which have been suggested as other investigations for HF in "ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012". Therefore, exercise testings will be applied upon physicians' need or judgment.

Firstly, this study is to assess the effect of AAIR pacing treatment for HF patients with CI in terms of exercise tolerance and quality of life. Specifically, the study will assess the changes in cardiac function associated with changes of physical exercise intensity and heart rate in AAIR pacing mode compared with AAI pacing mode. Secondly, the study will look at clinical outcomes in terms of NYHA class, 6MHW, blood BNP, Echo measurements following pacemaker therapy for 1 year. 6MHW and treadmill tests have been suggested as other investigations for HF in "ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012" and will be performed upon physicians' need or judgment.

The study will enroll up to 30 subjects that meet the indication for pacing therapy. Consented subjects will receive pacing therapy and two follow-ups in the following one year.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to give informed consent.
* Patient is between 18 and 70 years of age (including 18 and 70 years of age).
* Patients can perform treadmill exercise test for at least 8 minutes.
* Patient has been diagnosed with stable chronic HF according to HF guidance, including HFpEF (Heart Failure with preserved Ejection Fraction) and HFrEF (Heart Failure with reduced Ejection Fraction) patients.
* NYHA class I- III, with left ventricular ejection fraction less than 55% and more than 25%.
* Heart rate during treadmill test cannot reach 70% APMHR (Age Predicted Maximal Heart Rate) in (diagnostic criteria for CI, in accordance with class IA indications of pacing therapy for CI).

Exclusion Criteria:

* Patient with severe liver or kidney dysfunction.
* Patient has contraindications for pacing therapy.
* Patient has CI and is under appropriate clinical therapy.
* Patient has persistent or permanent atrial fibrillation (AF).
* Patient whose heart rate baseline at resting state is greater than 95 beats per minutes (BPM).
* Patient has contraindications for cardio-pulmonary exercise testing, including but not limited to unstable angina, decompensated heart failure, active pericarditis or myocarditis, hypertrophic cardiomyopathy, valvular heart disease and ECG ST-segment shift > 2mm at resting state.
* Less than 6 months after angina and ST dynamic changes during last 3 months.
* Patient with class I (with PR interval more than 200ms), II or III atrioventricular block, or interventricular block.
* NYHA Class IV.
* Less than 45 days after myocardial infarction.
* Less than 3 months after acute heart failure.
* Patient has uncontrolled hypertension.
* Patient is unwilling to sign the patient informed consent.
* Patient is pregnant or has pregnancy intention in the study duration.
* Patient has a medical condition that would limit study participation.
* Patient is enrolled in a concurrent study that may affect the outcome of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the study, total 30 heart failure patients with chronotropic incompetence who meet the inclusion and exclusion criteria would be enrolled from the ourtpatients in Fuwai Hospital.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-10-09 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
The treadmill walk duration change | The treadmill walk duration change from 3-6 months to 6-12 months post pacemaker implantation

SECONDARY OUTCOMES:
The 6 minutes hall walk distance change | 3-6 months and 6-12 months post pacemaker implantation

CONTACTS AND LOCATIONS:
Overall Officials: Shu Zhang, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No